CLINICAL TRIAL: NCT00397891
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Safety, Tolerability, and Pharmakokinetic Study of Single Ascending Doses of AAB-001 in Japanese Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Study Evaluating Single Ascending Doses of AAB-001 Vaccine SAD Japanese Patients With Alzheimers Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3133K1-102
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Results first posted 2014-09-04 (Estimated); Last update posted 2014-09-04 (Estimated); Status verified 2014-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — bapineuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): bapineuzumab 0.15 mg/kg or placebo
  Interventions: Drug: bapineuzumab
- 2 (Experimental): bapineuzumab 0.5 mg/kg or placebo
  Interventions: Drug: bapineuzumab
- 3 (Experimental): bapineuzumab 1.0 mg/kg or placebo
  Interventions: Drug: bapineuzumab

INTERVENTIONS:
Drug: bapineuzumab — The dose cohorts are as follows: 0.15 mg/kg AAB-001; 0.5 mg/kg AAB-001; 1.0 mg/kg AAB-001. Placebo is vehicle (all ingredients except active). In each dose cohort, designated as groups 1 to 3, study drug (AAB-001 or placebo) will be administered as an intravenous infusion over 1 hour.
  Arms: 1
Drug: bapineuzumab — The dose cohorts are as follows: 0.15 mg/kg AAB-001; 0.5 mg/kg AAB-001; 1.0 mg/kg AAB-001. Placebo is vehicle (all ingredients except active). In each dose cohort, designated as groups 1 to 3, study drug (AAB-001 or placebo) will be administered as an intravenous infusion over 1 hour.
  Arms: 2
Drug: bapineuzumab — The dose cohorts are as follows: 0.15 mg/kg AAB-001; 0.5 mg/kg AAB-001; 1.0 mg/kg AAB-001. Placebo is vehicle (all ingredients except active). In each dose cohort, designated as groups 1 to 3, study drug (AAB-001 or placebo) will be administered as an intravenous infusion over 1 hour.
  Arms: 3

SUMMARY:
Evaluate safety, tolerability, and pharmacokinetics of single doses of the investigational AAB-001 Vaccine in Japanese patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AD
* Age 50-85
* MMSE 14-26
* Other Inclusion Criteria Apply

Exclusion Criteria:

* Significant Neurological Disease
* Major Psychiatric Disorder
* Clinically Significant Systemic Illness
* Other Exclusion Criteria Apply

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- Japan (4):
  - Pfizer Investigational Site, Chiba
  - Pfizer Investigational Site, Saitama
  - Pfizer Investigational Site, Shizuoka
  - Pfizer Investigational Site, Tokyo

REFERENCES:
- [Derived] Arai H, Umemura K, Ichimiya Y, Iseki E, Eto K, Miyakawa K, Kirino E, Shibata N, Baba H, Tsuchiwata S. Safety and pharmacokinetics of bapineuzumab in a single ascending-dose study in Japanese patients with mild to moderate Alzheimer's disease. Geriatr Gerontol Int. 2016 May;16(5):644-50. doi: 10.1111/ggi.12516. Epub 2015 Jun 4. PMID 26044070
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=3133K1-102&StudyName=Study%20Evaluating%20Single%20Ascending%20Doses%20of%20AAB-001%20Vaccine%20SAD%20Japanese%20Patients%20With%20Alzheimers%20Disease

RESULTS

PARTICIPANT FLOW:
Groups:
- Bapineuzumab 0.15 mg/kg: Single dose of bapineuzumab (AAB-001) 0.15 milligram per kilogram (mg/kg) intravenous infusion over 1 hour on Day 1.
- Bapineuzumab 0.5 mg/kg: Single dose of bapineuzumab 0.5 mg/kg intravenous infusion over 1 hour on Day 1.
- Bapineuzumab 1.0 mg/kg: Single dose of bapineuzumab 1.0 mg/kg intravenous infusion over 1 hour on Day 1.
- Bapineuzumab 2.0 mg/kg: Single dose of bapineuzumab 2.0 mg/kg intravenous infusion over 1 hour on Day 1.
- Placebo: Single dose of placebo matched to bapineuzumab intravenous infusion over 1 hour on Day 1.
Period: Overall Study
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 8
Completed | 5 | 6 | 6 | 6 | 7
Not Completed | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.67 (5.16) | 72.17 (8.38) | 72.17 (10.87) | 64.83 (5.19) | 68.75 (8.89) | 67.78 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 3 | 3 | 4 | 14
  Male | 3 | 5 | 3 | 3 | 4 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study medication without regard to possibility of causal relationship. SAE: an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between dose of study medication and up to 52 weeks after the dose that were absent before treatment or that worsened relative to pre-treatment state.
Time Frame: Baseline up to Week 52
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants
  AEs | 5 | 3 | 6 | 3 | 7
  SAEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examination included the assessment of abdomen, back/spinal, breasts, external genitalia, extremities, general appearance, head, eyes, ears, nose, throat (HEENT), heart, lungs, lymph nodes and skin.
Time Frame: Screening up to Week 52
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Signs of Potential Clinical Importance
Description: Criteria for determining potentially clinically important (PCI) vital signs was described as: supine blood pressure (BP)- systolic (greater than or equal to [>=]160 millimeter mercury [mm Hg] or less than or equal to [<=]90 mm Hg and increase or decrease of >=20 mm Hg compared to baseline value), supine diastolic BP (>=100 mm Hg or <= 50 mm Hg and increase or decrease of >=15 mm Hg compared to baseline value), supine pulse rate (>=120 beats per minute (bpm) or <=45 bpm and increase or decrease of >15 bpm compared to baseline value), body temperature (>38.3 degree Celsius and <35 degree Celsius).
Time Frame: Baseline up to Week 52
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 2 | 0 | 2 | 1 | 1

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Results of Potential Clinical Importance
Description: Criteria for determining PCI ECG result was described as: heart rate (>=120 bpm or <=45 bpm and increase or decrease of >15 bpm compared to baseline value), PR interval (>=220 millisecond (msec) and change of >=20 msec compared to baseline value), QRS interval (>=120 msec), corrected QT (QTc) interval for men (>450 msec), QTc interval for women (>470 msec).
Time Frame: Screening up to Week 16
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 1

5. Primary Outcome: Number of Participants With Laboratory Test Results of Potential Clinical Importance
Description: Criteria for PCI laboratory results: hematology (hematocrit [decrease >=5%], hemoglobin [decrease >=20gram/liter {g/L}] from baseline, white blood cells [<3], neutrophils [<1.5], platelet [<100], eosinophils [>0.5] *10^9/L); blood chemistry (sodium [>5], potassium [>0.5], fasting glucose [>0.83], phosphorous [>0.162] millimole/L [mmol/L] above upper limit of normal [ULN] and below lower limit of normal [LLN], non-fasting glucose >5 mmol/L above ULN, >0.56 mmol/L below LLN, creatinine >1.36*ULN, blood urea nitrogen >1.5*ULN, calcium [change of >=0.25 mmol/L], total protein [change of >=20g/L], albumin [change of >=10g/L], uric acid [change of >0.119mmol/L] from baseline and outside normal limits); Liver function tests (alanine aminotransferase/serum glutamic pyruvic transaminase [ALT/SGPT] and aspartate aminotransferase/serum glutamic oxaloacetic transaminase [AST/SGOT] >2*ULN, total bilirubin >2*ULN, alkaline phosphatase >1.5*ULN, gamma-glutamyl-transpeptidase [GGT] >3*ULN).
Time Frame: Week 1 up to Week 52
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 6 | 4 | 3 | 5 | 5

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Neurological Examinations
Description: Neurological examination included the assessment of mental status, cranial nerves, visual fields, sensory, motor, gait, primitive reflexes and tendon reflexes.
Time Frame: Screening up to Week 52
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Score at Week 6
Description: MMSE measures general cognitive functioning: orientation to time (range: 0 to 5) and orientation to place (range: 0 to 5), registration of 3 words (range: 0 to 3), attention and calculation (range: 0 to 5), recall of 3 words (range: 0 to 3), naming (range: 0 to 2), repetition (range: 0 to 1), comprehension (range: 0 to 3), reading (range: 0 to 1), writing (range: 0 to 1) and drawing (range: 0 to 1). Total score is the sum of sub-scores; total score ranges from 0 to 30, higher score indicates better cognitive state.
Time Frame: Baseline, Week 6
Population: Safety data set included all randomized participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
units on a scale
  Baseline | 16.8 (2.9) | 21.0 (3.6) | 21.0 (4.6) | 20.2 (2.8) | 20.6 (3.0)
  Change at Week 6 | -0.2 (2.1) | 0.0 (2.3) | -0.3 (3.0) | -0.2 (3.8) | -1.9 (3.1)

8. Primary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Score at Week 16
Description: as for outcome 7
Time Frame: Baseline, Week 16
Population: Safety data set included all randomized participants who received at least 1 dose of study medication. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 7
units on a scale | 0.2 (2.9) | -0.7 (4.1) | 0.7 (2.4) | -0.3 (2.4) | -1.4 (2.6)

9. Primary Outcome: Change From Baseline in Mini-Mental State Examination (MMSE) Score at Week 52
Description: as for outcome 7
Time Frame: Baseline, Week 52
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 7
units on a scale | -2.4 (1.9) | -3.8 (6.4) | -0.7 (2.7) | -1.2 (5.6) | -2.9 (1.3)

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Bapineuzumab
Description: Participants who received bapineuzumab were reported.
Time Frame: 0 (pre-infusion), 0.5, 1, 1.5, 2, 4, 6 hours post start of infusion on Day 1; Day 2, 3; Week 1, 2, 4, 6, 8, 11, 13, 16, 26, 52
Population: Pharmacokinetic (PK) data set included all randomized participants who had at least 1 available data of serum bapineuzumab, serum anti-bapineuzumab antibody or plasma amyloid beta concentration.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
microgram per milliliter (mcg/mL) | 3.32 (0.857) | 11.1 (1.16) | 21.0 (0.968) | 61.0 (32.8)

11. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of Bapineuzumab
Description: Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: PK data set included all randomized participants who had at least 1 available data of serum bapineuzumab, serum anti-bapineuzumab antibody or plasma amyloid beta concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 1.51 [1.08 to 3.91] | 1.54 [1.00 to 5.86] | 1.53 [1.00 to 2.00] | 1.71 [0.45 to 5.95]

12. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration [AUC (0-t)] of Bapineuzumab
Description: AUC is a measure of the serum concentration of the drug over time. AUC (0-t) is area under the serum concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t). Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg*hour/mL
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg*hour/mL | 1260 (254) | 4264 (462) | 7818 (652) | 15313 (8478)

13. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0 - ∞)] of Bapineuzumab
Description: AUC is a measure of the serum concentration of the drug over time. AUC (0 - ∞) is area under the serum concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - ∞). It is obtained from AUC (0 - t) plus AUC (t - ∞). Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mcg*hour/mL
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mcg*hour/mL | 1279 (266) | 4323 (456) | 7884 (640) | 15405 (8438)

14. Secondary Outcome: Systemic Clearance (CL) of Bapineuzumab
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL/hour | 6.88 (1.32) | 7.49 (1.71) | 7.23 (1.49) | 8.84 (3.97)

15. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Bapineuzumab
Description: Volume of distribution is defined as the theoretical blood volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Steady state volume of distribution (Vss) is the apparent volume of distribution at steady-state. Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
mL | 5574 (906.5) | 5947 (1406) | 5827 (1611) | 6879 (3132)

16. Secondary Outcome: Mean Residence Time of Bapineuzumab
Description: MRT is average time for which the drug molecules resides in the body, after administration. It is calculated as area under the serum concentration versus time first moment curve from time zero (pre-dose) to extrapolated infinite time (AUMC [0 - ∞]) divided by area under the plasma concentration versus time curve from time zero (pre-dose) to extrapolated infinite time (AUC[0 - ∞]). AUMC (0-∞) is calculated as AUMC(0-inf)= AUMCt + [(t x Ct) / kel] + (Ct / kel^2). AUMCt is the area under the first moment curve from zero time to time t calculated using the trapezoidal method, Ct is the concentration at time t and kel is the terminal phase rate constant. Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
days | 34.5 (7.0) | 33.3 (4.4) | 33.4 (5.2) | 32.4 (4.6)

17. Secondary Outcome: Serum Decay Half-Life (t1/2) of Bapineuzumab
Description: Serum decay half-life is the time measured for the serum concentration to decrease by one half. Participants who received bapineuzumab were reported.
Time Frame: as for outcome 10
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
days | 28.1 (5.9) | 26.7 (1.8) | 26.2 (3.4) | 15.0 (9.9)

18. Secondary Outcome: Serum Bapineuzumab Concentrations
Description: Serum bapineuzumab concentration was determined by using a validated enzyme-linked immunosorbent assay (ELISA) method. Participants who received bapineuzumab were reported.
Time Frame: 0 (pre-infusion), 0.5, 1, 1.5, 2, 4, 6, 24, 48, 168, 336, 672, 1008, 1344, 1848, 2184, 2688, 4368, 8736 hours post start of infusion
Population: PK data set included all randomized participants who had at least 1 available data of serum bapineuzumab, serum anti-bapineuzumab antibody or plasma amyloid beta concentration. Here 'n' signifies those participants who were evaluable for this measure at the specified time point for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per milliliter (ng/mL)
  0 Hour (n=0,0,0,0) | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable.
  0.5 Hour (n=6,5,6,6) | 1602 (464) | 5211 (1025) | 8158 (332) | 29206 (26241)
  1 Hour (n=6,6,6,6) | 2970 (624) | 10259 (1421) | 19939 (868) | 48995 (41719)
  1.5 Hour (n=6,6,6,6) | 3093 (696) | 10861 (1398) | 20423 (1559) | 43798 (34612)
  2 Hour (n=6,6,6,6) | 2854 (726) | 10362 (1473) | 19200 (1333) | 48008 (26387)
  4 Hour (n=6,6,6,6) | 2917 (1079) | 10044 (1564) | 17588 (1762) | 32399 (14264)
  6 Hour (n=6,6,6,6) | 2678 (845) | 9753 (1209) | 18935 (1194) | 34349 (14934)
  24 Hour (n=6,6,6,6) | 2276 (665) | 7774 (1249) | 12983 (224) | 25567 (20599)
  48 Hour (n=6,6,6,6) | 1946 (379) | 6423 (774) | 12179 (372) | 20575 (18648)
  168 Hour (n=6,6,6,6) | 1279 (225) | 4431 (826) | 8170 (369) | 15925 (10963)
  336 Hour (n=6,6,6,6) | 911 (271) | 3441 (344) | 6374 (547) | 12325 (5331)
  672 Hour (n=6,6,6,6) | 599 (80) | 1940 (328) | 3379 (1409) | 6720 (4830)
  1008 Hour (n=6,6,6,6) | 384 (127) | 1396 (326) | 2295 (376) | 5064 (2197)
  1344 Hour (n=6,6,6,6) | 267 (76) | 811 (120) | 1389 (318) | 4440 (1755)
  1848 Hour (n=6,6,6,6) | 158 (61) | 519 (126) | 990 (312) | 2172 (1289)
  2184 Hour (n=6,6,4,6) | 107 (49) | 375 (95) | 796 (126) | 1386 (950)
  2688 Hour (n=6,6,6,6) | 69 (41) | 221 (96) | 468 (101) | 595 (678)
  4368 Hour (n=5,5,6,2) | 14 (12) | 46 (20) | 70 (28) | 25 (10)
  8736 Hour (n=0,0,0,0) | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable. | NA (NA) — Concentration was not estimable since no participant was evaluable.

19. Secondary Outcome: Number of Participants With Positive Serum Anti-Bapineuzumab Antibody
Description: Serum anti-bapineuzumab antibody concentration was determined by using a validated ELISA method.
Time Frame: Baseline (Day 1) up to Week 52
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Plasma Amyloid-beta (x-40) Concentrations
Description: Amyloid-beta (A-beta) is a peptide fragment of the amyloid precursor protein which is one of the characteristic hallmarks of Alzheimer's disease (AD). Total plasma amyloid-beta (x-40) was determined using a validated ELISA method.
Time Frame: 0 (pre-infusion), 1, 6, 24, 336, 1008, 2184, 2688, 4368, 8736 hours post start of infusion
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: picogram per milliliter (pg/mL)
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
picogram per milliliter (pg/mL)
  0 Hour (n=6,6,6,6,8) | 309 (116) | 298 (91) | 276 (43) | 339 (20) | 281 (38)
  1 Hour (n=6,5,5,6,8) | 1009 (369) | 1050 (142) | 1593 (88) | 1708 (247) | 292 (48)
  6 Hour (n=6,6,6,6,8) | 1697 (871) | 2664 (509) | 3755 (356) | 3905 (656) | 293 (40)
  24 Hour (n=6,6,6,6,8) | 1474 (844) | 3581 (660) | 5333 (426) | 7405 (1630) | 302 (71)
  336 Hour (n=6,6,6,6,8) | 784 (320) | 1675 (396) | 3345 (485) | 4325 (670) | 279 (54)
  1008 Hour (n=6,6,6,6,8) | 543 (219) | 985 (328) | 1566 (281) | 2664 (601) | 287 (41)
  2184 Hour (n=6,6,6,6,7) | 331 (119) | 488 (142) | 668 (157) | 1149 (432) | 278 (59)
  2688 Hour (n=6,6,6,6,7) | 341 (108) | 471 (114) | 528 (128) | 803 (268) | 307 (81)
  4368 Hour (n=5,6,6,6,7) | 302 (86) | 310 (74) | 351 (33) | 425 (68) | 291 (71)
  8736 Hour (n=5,6,6,6,7) | 298 (107) | 308 (29) | 342 (41) | 299 (22) | 283 (42)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Bapineuzumab 0.15 mg/kg | Bapineuzumab 0.5 mg/kg | Bapineuzumab 1.0 mg/kg | Bapineuzumab 2.0 mg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 5/6 | 3/6 | 6/6 | 3/6 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bapineuzumab 0.15 mg/kg (N=6) | Bapineuzumab 0.5 mg/kg (N=6) | Bapineuzumab 1.0 mg/kg (N=6) | Bapineuzumab 2.0 mg/kg (N=6) | Placebo (N=8)
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 1
Glaucoma (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Injection site haemorrhage (General disorders) | 1 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpangina (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 2
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0
Tinea infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Nystagmus (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Parkinsonism (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.